CLINICAL TRIAL: NCT06646510
Title: Effect of Sensory Electrical Stimulation on Resting Tremors in Patients with Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Yassen, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005124
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): traditional treatment of hand tremors
  Interventions: Other: traditional exercises
- study group (Experimental): traditional treatment in addition to sensory electrical stimulation
  Interventions: Other: traditional exercises; Other: sensory electrical stimulation

INTERVENTIONS:
Other: traditional exercises — strengthening exercise for the shoulder muscles( shoulder extensors, shoulder retractors from prone position and shoulder external rotation exercise for 3 sets 10 repetition , weight bearing exercise on the hand from quadruped position and sitting position and strengthening exercise on the intrinsic muscles of the hand
Other: sensory electrical stimulation — The stimulated muscles included the flexor carpi radialis (FCR), extensor carpi radialis (ECR), and flexor carpi ulnaris (FCU). Rectangular surface electrodes (Ag/AgCl; 50mm _ 50mm size) were attached on the motor point of each muscle, i.e., at four fingerbreadths from biceps tendon of FCR, at two fingerbreadths distal from lateral epicondyle for the ECR, at two fingerbreadths volar to ulna at the junction of the upper and middle thirds of the forearm for FCU.14 Portable stimulators will use with the following stimulation settings: constant current (0.2 mA step), 100 Hz stimulation frequency, biphasic pulse, and 300 _s pulsewidth.
  Arms: study group

SUMMARY:
Parkinson's disease is one of the most prevalent motor disorders in the world . The disease is progressive and has no known treatment. In addition to a number of psychological and autonomic issues, the disease also cause movement abnormalities which are the most challenging problem because management is still limited by medication or traditional physiotherapy the most effective way to treat symptoms is through an interprofessional new modalities as sensory stimulation , this study will be the first of its type to measure the effect of sensory stimulation on static tremors. Also, this study is the first of its type to make a continues treatment protocol for patient with static tremors.

SO the purpose of these study will To investigate the effect of sensory electrical stimulation on resting tremors in Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 60
* Diagnosed with idiopathic Parkinson's disease with Magnetic resonance imaging of the brain
* All the patients will have mild to moderate symptoms based on (the Unified Parkinson's Disease Rating Scale UPDRS) ≥ 3
* Static tremors have been present at the hand and wrist
* Absence of other disorders that cause similar symptoms like dystonia

Exclusion Criteria:

* History of hand trauma causes stiffness
* Presence of other neurological problems interferes with diagnosis as hemiplegic stroke
* Secondary parkinsonism (drug-induced or vascular ) which has very low tremor magnitude which can not be detected The patient has a severe visual problem that does not allow following the instructions.
* The patient educational level does not allow for following the instructions.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-05 (Estimated)

PRIMARY OUTCOMES:
triaxial gyrosensor (accelerator) | 3 weeks
  Three-dimensional angular motion will measured at the index finger of the more affected hand, by using triaxial gyrosensor (STM32L151, STMicroelectronics, ). The gyrosensor will embedded in an elastic band and attached on the dorsum of proximal phalanx
Fahn-tolosa- marin clinical rating scale | 3 weeks
  Fahn_tolosa_marin clinical rating scale( FTM) is avalid scale for asses hand tremor, it consist of two items related to the hand , 1_trmors 2_hand writing The score is form 0 to 4 , 0 mean no tremors , 4 means severe tremors

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinics, Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided